CLINICAL TRIAL: NCT05406999
Title: A Prospective, Multi-arm, Multi-center Clinical Trial on Neoadjuvant Intense Endocrine Therapy for High Risk and Locally Advanced Prostate Cancer
Brief Title: Neoadjuvant Intense Endocrine Therapy for High Risk and Locally Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-118
Record Dates: First submitted 2022-05-29; First posted 2022-06-07 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Neoadjuvant Therapy; High Risk Prostate Cancer; Locally Advanced Prostate Cancer; Intense Endocrine Therapy
MeSH Terms: interventions — Abiraterone Acetate; Prednisolone; enzalutamide; apalutamide; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- ADT alone + prostatectomy (Active Comparator): A total of 100 subjects receive ADT for 6 cycles (28 days per cycle) before prostatectomy. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Procedure: Robot-assisted radical prostatectomy
- ADT plus Abiraterone (Experimental): A total of 150 subjects in this group received abiraterone acetate + prednisolone acetate daily for 6 cycles along with ADT. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Drug: Abiraterone Acetate; Drug: Prednisolone tablets; Procedure: Robot-assisted radical prostatectomy
- ADT plus Enzalutamide (Experimental): A total of 50 subjects in this group received enzalutamide daily for 6 cycles along with ADT. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Drug: Enzalutamide; Procedure: Robot-assisted radical prostatectomy
- ADT plus Apalutamide (Experimental): A total of 150 subjects in this group received apalutamide daily for 6 cycles along with ADT. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Drug: Apalutamide; Procedure: Robot-assisted radical prostatectomy
- ADT plus Darotamide (Experimental): A total of 150 subjects in this group received darotamide daily for 6 cycles along with ADT. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Drug: Darotamide; Procedure: Robot-assisted radical prostatectomy
- ADT plus Rizvilutamide (Experimental): A total of 150 subjects in this group received rizvilutamide daily for 6 cycles along with ADT. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Drug: Rezvilutamide; Procedure: Robot-assisted radical prostatectomy
- PARP inhibitor + abiraterone + ADT (Experimental): A total of 100 subjects in this group received Poly ADP-ribose Polymerase (PARP) Inhibitor plus abiraterone along with ADT. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Drug: Abiraterone Acetate; Drug: Prednisolone tablets; Drug: PARP inhibitor; Procedure: Robot-assisted radical prostatectomy
- PARP inhibitor + ADT (Experimental): A total of 50 subjects in this group in this group received Poly ADP-ribose Polymerase (PARP) Inhibitor along with ADT mentioned above. Enrolled patients carry homologous recombination repair (HRR) gene mutation verified by molecular testing. Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.
  Interventions: Drug: ADT; Drug: PARP inhibitor; Procedure: Robot-assisted radical prostatectomy

INTERVENTIONS:
Drug: ADT — The ADT regimen will be determined by the investigators at separate centers. The dose and frequency of administration will be consistent with the prescribing information. Available drugs include triptorelin, goserelin, leuprolide, digareke ect.
Drug: Abiraterone Acetate — 1000 mg (250 mg×4 tablets) once daily, orally
  Arms: ADT plus Abiraterone; PARP inhibitor + abiraterone + ADT
Drug: Prednisolone tablets — 5 mg once daily, orally.
  Arms: ADT plus Abiraterone; PARP inhibitor + abiraterone + ADT
Drug: Enzalutamide — 160 mg (40 mg× 4 tablets) once daily, orally.
  Arms: ADT plus Enzalutamide
Drug: Apalutamide — 240 mg (60 mg×4 tablets) once daily, orally.
  Arms: ADT plus Apalutamide
Drug: Darotamide — 600 mg (300 mg × 2 tablets) twice daily, orally.
  Arms: ADT plus Darotamide
Drug: Rezvilutamide — 240 mg (80 mg × 3 tablets) once daily orally
  Arms: ADT plus Rizvilutamide
Drug: PARP inhibitor — The PARP inhibitors will be determined by the investigators at separate centers. The dosage and frequency of administration will be consistent with the prescribing information. Available drugs include olaparib, fluzoparib, pamiparib, talazoparib ect.
  Arms: PARP inhibitor + ADT; PARP inhibitor + abiraterone + ADT
Procedure: Robot-assisted radical prostatectomy — Robot-assisted radical prostatectomy was performed within 2 weeks after the end of the therapy.

SUMMARY:
This is a prospective, multicenter, multi-arm, non-randomized, open-label clinical trial to evaluate the efficacy and safety of neoadjuvant intense endocrine therapy for high-risk or locally advanced prostate cancer.

DETAILED DESCRIPTION:
The study was designed to evaluate the efficacy and safety of different forms of neoadjuvant intense androgen deprivation therapy (ADT) compared with ADT alone, followed by prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have been histologically diagnosed of prostate cancer and must be eligible for radical prostatectomy.
2. All patients must undergo thorough tumor staging and meet one of the following criteria: a) multi-parameter MRI or PSMA PET/CT shows clinical staging of primary tumor ≥ T3; b) Gleason score of primary tumor ≥ 8; c)prostate specific antigen(PSA) ≥20 ng/ml; d) Imaging evaluation shows regional lymph node metastases (N1).
3. Eastern Cooperative Oncology Group (ECOG) physical condition score ≤ 1.
4. Patients must have adequate hematologic function, hepatic function, renal function and cardiac function.
5. Patients must participate voluntarily and sign an informed consent form(ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must bewilling to obey the prohibitions and restrictions specified in the research protocol.
6. Fertile patients must be willing to use highly effective contraception during the study period and within 120 days of the last dose of treatment.

Exclusion Criteria:

1. Patients with neuroendocrine, small cell, or sarcoma-like pathologic features are not eligible.
2. Patients with low-risk or medium-risk, localized prostate cancer (the following conditions are met at the same time) are not eligible: a) multiparameter MRI or PSMA PET / CT shows clinical staging of primary tumor < T3; b) Gleason score of primary tumor < 8; c) prostate specific antigen (PSA) <20 ng/ml.
3. Patients with clinical or radiological evidence of extra-regional lymph node metastases or bone metastases or visceral metastases (any M1) are not eligible.
4. Patients who have previously received androgen deprivation therapy (medical or surgical) or focal treatment, radiotherapy, chemotherapy for prostate cancer are not eligible.
5. Patients with severe or uncontrolled concurrent infections are not eligible.
6. Patients must not have New York Heart Association Class III or IV congestive heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction within 6 months prior to registration.
7. Patients must not have uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
8. Patients must not have had other malignancies other than prostate cancer in the past 5 years, but cured basal cell or squamous cell skin cancers can be enrolled.
9. Patients with mental illness, mental disability or inability to give informed consent are not eligible.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate | up to 3 years
  Pathologic response rate= Pathologic Complete Response (pCR) Rate + Minimal Residual Disease (MRD) rate
3 year biochemical progression free survival (bPFS) | up to 3 years
  Biochemical progression free survival (bPFS) within 3 years

SECONDARY OUTCOMES:
Metastasis-Free Survival (MFS) | up to 5 years
  Metastasis-Free Survival (MFS) after intense neoadjuvant therapy
Time to castration-resistant prostate cancer（CRPC) | up to 5 years
  Time to castration-resistant prostate cancer（CRPC) after intense neoadjuvant therapy
PSA response rate | up to 3 years
  Prostate specific antigen (PSA) drops ≥ 98% after intense neoadjuvant therapy
Positive margin rate | up to 6 months
  The positive margin rate of whole-mount pathology for prostatectomy after intense neoadjuvant therapy
Pathologic downgrade rate | up to 6 months
  The pathologic downgrade rate of whole-mount pathology for prostatectomy after intense neoadjuvant therapy compared with initial T stage.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. All grades of adverse events will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No